CLINICAL TRIAL: NCT01514591
Title: Thromboelastography to Assess Hemostatic Changes in Laboring Patients Undergoing Non-elective (Intrapartum) Cesarean Delivery
Brief Title: Thromboelastography in Non-elective Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alex James Butwick, Principal Investigator, Stanford University
Other Study IDs: SU-08162011-8270; IRB 22205 (Other: Stanford IRB)
Record Dates: First submitted 2012-01-11; First posted 2012-01-23 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for TEG analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Non-elective Cesarean Delivery: We will only enroll patients undergoing non-elective CS with an 'epidural top-up' for surgical anesthesia. By definition, our study will only apply to laboring women with working labor epidurals (which were provided for labor analgesia).

SUMMARY:
The purpose of the study is to assess the coagulation changes that occur in laboring patients undergoing non-elective (intrapartum)Cesarean delivery using thromboelastography (TEG). We will compare coagulation data to assess potential coagulation changes associated with hemoglobin changes before and after surgery, and related to estimated blood loss.

DETAILED DESCRIPTION:
The purpose of the study is to assess the coagulation changes that occur in laboring patients undergoing non-elective (intrapartum)Cesarean delivery using thromboelastography (TEG). TEG is a point- of-care device which measures the viscoelastic properties of clot formation. This device can provide rapid and detailed information about coagulation changes in the perioperative period. We will compare coagulation data collected from the study to assess potential coagulation changes associated with Hemoglobin changes before and after surgery, and related to estimated blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric in-patients
* Laboring patients with Epidurals for Labor Analgesia going for non-elective Cesarean
* Patients of all ethnic backgrounds will be included
* Singleton pregnancy
* ASA 1 or 2

Exclusion Criteria:

* Patients with underlying coagulation disorders.
* Patients with thrombocytopenia (platelet count <100).
* Patients with pregnancy-induced hypertension, pre-eclampsia.
* Patients requiring the following medications prior to surgery: NSAIDS, aspirin, anticoagulants.
* Patients requiring elective Cesarean delivery.
* Patients with significant obstetric or medical disease.
* No patients <18 years of age will be recruited.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obstetrical laboring patients who are undergoing non-elective Cesarean delivery with an 'epidural top up' for surgical anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss; Coagulation data (Thromboelastography, Laboratory) | pre and post cesarean delivery, an expected average of 75 minutes
  This study will allow us to collect more information about the hemostatic effects that occur during non-elective Cesarean delivery. This information will add to current knowledge base (which we have published) about coagulation changes in the peripartum period in patients undergoing non-elective Cesarean section.

SECONDARY OUTCOMES:
Hematologic indices | Pre and post cesarean delivery, an expected average of 75 minutes
  Hematologic indices will include: Hemoglobin concentration and platelet count.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Butwick, MBBS, FRCA, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Stanford, California, United States

REFERENCES:
- [Background] Butwick A, Ting V, Ralls LA, Harter S, Riley E. The association between thromboelastographic parameters and total estimated blood loss in patients undergoing elective cesarean delivery. Anesth Analg. 2011 May;112(5):1041-7. doi: 10.1213/ANE.0b013e318210fc64. Epub 2011 Apr 7. PMID 21474664